CLINICAL TRIAL: NCT05858775
Title: MAPVIX: Mapping the Uterine Cervix Stiffness of Pregnant Women at Mid Gestation
Brief Title: Mapping the Uterine Cervix Stiffness of Pregnant Women at Mid Gestation
Acronym: MAPVIX
Status: Completed | Type: Observational
Sponsor: Pregnolia AG (Industry)
Responsible Party: Sponsor
Other Study IDs: F-405-11 v. 2.0, 2023-02-1
Record Dates: First submitted 2023-05-03; First posted 2023-05-15 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Cervix; Pregnancy
Keywords: Cervical Stiffness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Nulliparous cohort: Nulliparous pregnant woman
  Interventions: Device: Pregnolia System
- Multiparous cohort: Multiparous pregnant woman
  Interventions: Device: Pregnolia System

INTERVENTIONS:
Device: Pregnolia System — Cervical stiffness assessment with the Pregnolia System at 3 locations on the uterine cervix.

SUMMARY:
The assessment of cervical stiffness plays a major role in obstetrics, for example to assess the risk of preterm birth.

The Pregnolia System is a CE-certified measuring device that objectively determines cervical stiffness using a slight negative pressure. The Pregnolia System was developed in Switzerland and resulted from a research project of the ETH and the University Hospital Zurich.

Until now, the stiffness of the cervix was examined and individually assessed by palpation (palpation with fingers). The Pregnolia System was developed to make this measurement objective and independent of the examining person.

The aim of the study is to measure cervical stiffness at different locations on the cervix to see if there are differences between the measurement locations.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent signed by the subject
* Pregnant woman at GA 16+0 - 22+6
* Singleton pregnancy
* 18 years or older
* Nulliparous cohort: nulliparous pregnant woman
* Multiparous cohort: multiparous pregnant woman

Exclusion Criteria:

* Lack of informed consent
* Placenta praevia
* Severe vaginal bleeding
* Rupture of membranes before 34 weeks (to be excluded with pH test)
* Visible tissue scarring at the measurement locations* on cervix
* Light bleeding (if the bleeding can be stopped, it is no longer an exclusion criterion)
* Cervical dilation ≥ 3 cm
* Cerclage or pessary in place
* Vaginal or cervical infections (to be excluded with the Amsel criteria)

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant women at gestational ages between 16+0 - 22+6 weeks
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2023-07-05 (Actual); Primary Completion 2025-10-10 (Actual); Study Completion 2025-10-10 (Actual)

PRIMARY OUTCOMES:
Cervical Stiffness Index at 16+0 - 22+6 | 16+0 - 22+6 gestational weeks
  Cervical Stiffness Index (CSI, in mbar) measured at 3 locations on the cervix (approximately 12, 4 and 8 o'clock, in a random order) at mid-pregnancy (16+0 - 22+6 gestational weeks).

SECONDARY OUTCOMES:
Cervical Stiffness Index (repetition) | 16+0 - 22+6 gestational weeks and optional follow-up visits
  Cervical Stiffness Index (CSI, in mbar) measured 3 times at each location
Cervical Stiffness Index (cohort) | 16+0 - 22+6 gestational weeks and optional follow-up visits
  Cervical Stiffness Index (CSI, in mbar) for each cohort.
Delivery data | 1-4 weeks after delivery or termination of the pregnancy
  Delivery data

CONTACTS AND LOCATIONS:
Locations (2):
- Switzerland (2):
  - gynosense AG, Uster
  - University Hospital Zurich, Zurich

IPD SHARING:
Plan to Share IPD: Undecided